CLINICAL TRIAL: NCT04995198
Title: PROMISE Registry: A Prostate Cancer Registry of Outcomes and Germline Mutations for Improved Survival and Treatment Effectiveness
Status: Recruiting | Type: Observational
Sponsor: Prostate Cancer Clinical Trials Consortium (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Fred Hutchinson Cancer Center (Other); Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other); Advancing Cancer Treatment, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: c19-235
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Genetics; Registry; Germline Mutation; Genetic Testing; Germline Testing
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Saliva, Blood (optional), Tissue (optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with at least one germline pathogenic/likely pathogenic variant
- Participants with at least one variant of uncertain significance

SUMMARY:
PROMISE aims to create a comprehensive nationwide registry of prostate cancer patients with germline pathogenic variants by prospectively screening approximately 5,000 subjects with a confirmed prostate cancer diagnosis, either through tissue biopsy, PSA greater than 100 ng/dL and/or radiographic evidence of disease and receiving systemic therapy for prostate cancer. Patients at all stages of disease will be welcome to participate in the PROMISE Registry.

Participants will be recruited & screened over a five-year period. Study participants will be asked to provide a saliva sample to be tested for germline cancer risk variants through Color Health. If the results identify a pathogenic or likely pathogenic variant, an appointment with a genetic counselor from Color Health will be scheduled to discuss the results.

Participants will complete a baseline demographic survey that includes self-reported health history, family history of cancer and standardized patient reported outcome (PRO) measures.

PROMISE Registry staff will request medical records from the participant's cancer care provider(s) for the purpose of obtaining clinical data.

Participants will receive bi-annual newsletters offering information on new developments in treatment and research opportunities, including clinical trials, associated with genetic variants.

Eligible participants (those with target germline mutations) will be followed every 6 months to obtain updated health records data and patient-reported outcomes data. Participants will be followed for a minimum of 15 years.

The PROMISE registry will help identify prostate cancer patients with pathogenic variants to learn more about how these variants affect patient outcomes. Ultimately, we hope to help patients learn more about their disease and the treatments that they may derive the most benefit from, including the germline genetic biomarker-based clinical trials they may be eligible for.

For more information, visit the study website at: prostatecancerpromise.org

ELIGIBILITY:
Inclusion Criteria:

* Have prostate cancer (any stage of disease or survivorship) diagnosed or documented through one of the following:

  * tissue biopsy, and/or
  * PSA greater than 100 ng/dL (1ng/ml), and/or
  * clear radiographic evidence of disease
* Live in the United States (including Puerto Rico, Guam, American Samoa, US Virgin Islands, Northern Mariana Islands)

Exclusion Criteria:

* Unable or unwilling to provide all of the necessary information for eligibility
* Incomplete inclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with prostate cancer (any stage of disease or survivorship). Individuals are eligible whether they have had prior germline genetic testing or not.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2036-02-26 (Estimated)

PRIMARY OUTCOMES:
Frequency of at least one germline pathogenic or likely pathogenic variant | 5 years
  Frequency of having at least one germline pathogenic or likely pathogenic variant in a cancer risk gene based on the number of subjects screened.

SECONDARY OUTCOMES:
Frequency of pathogenic or likely pathogenic germline variants of interest | 5 years
  Frequency of pathogenic or likely pathogenic germline variants of interest in subjects with prostate cancer. We will estimate the frequency of having each of the germline pathogenic or likely pathogenic variant in the cancer risk genes based on the number of subjects screened in each subpopulation.
Identify and recruit control group of patients with a variant of uncertain significance (VUS) | 5 years
  Identify and recruit a control group of patients with a VUS in their clinical or research results in the following genes: ATM, ATR, BARD1, BRCA1, BRCA2, FAM175A, GEN1, HOXB13, MRE11A, PALB2 and XRCC2.
Association between disease characteristics and genetic variants | 15 years
  Collect data on disease characteristics and examine the association between disease characteristics and pathogenic and likely pathogenic germline variants and VUS of interest.
Analysis of patient reported outcomes (PRO) measures | 15 years
  Collect PRO measures associated with genetic testing in subjects with prostate cancer using the validated EORTC QLQ-C30.
Analysis of longitudinal outcome data | 15 years
  Collect longitudinal outcome data on subjects with pathogenic and likely pathogenic germline variants and VUS of interest, for specific treatments, treatment sequences or therapy combinations used for treating prostate cancer.
Comparison of overall survival | 15 years
  Compare overall survival in subjects with pathogenic and likely pathogenic germline variants of interest and subjects with VUS.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Cheng, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Channing Paller, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (3):
- United States (3):
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PROMISE Study Site — http://www.prostatecancerpromise.org/